CLINICAL TRIAL: NCT04550429
Title: The Effect of Decreased Uterine Filling Pressure in Hysteroscopy, a Double-blind Control Trial
Brief Title: Uterine Filling Pressure in Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Professor of Obstetrics and Gynecology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STU00211845
Record Dates: First submitted 2020-08-28; First posted 2020-09-16 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Intervention Model Description: Using block randomization to divide patients into two groups using two different levels of pressure on the hysteroscopic morcellator: experimental group (those receiving 60 mmHg of pressure) and control group (those receiving 80 mmHg of pressure)
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 60 mmHg MyoSure Hysteroscopic Morcellator Device (Active Comparator): The rationale for this experimental arm is that the pressurization can result in excess fluid being absorbed by the patient without a substantial benefit to surgical outcome. Minimizing the pressure from 80 mmHg (which is standard of care) to 60 mmHg used during this procedure may optimize outcome without compromising visualization of the surgeon. The research procedure will take place in the operating room of the minimally invasive gynecologic surgery department.
  Interventions: Device: MyoSure Hysteroscopic Morcellator Device
- 80 mmHg MyoSure Hysteroscopic Morcellator Device (Sham Comparator): This is the standard of care pressurization for this procedure at Northwestern Medicine and will be the control group for the study
  Interventions: Device: MyoSure Hysteroscopic Morcellator Device

INTERVENTIONS:
Device: MyoSure Hysteroscopic Morcellator Device — This device is normally used for this procedure, but I included it as intervention because we will lower the pressure for one arm of the study (treatment) and keep the pressure in the other arm (control) as the standard of care.

SUMMARY:
The aim of the study is to compare the outcomes of patients undergoing hysteroscopy with a Myosure device with a pressure of 60 mmHg to those using the standard of 80 mmHg.

DETAILED DESCRIPTION:
An a priori sample size calculation was completed. To achieve 80% power and an alpha of .05, the study team needed a sample size of 68 total with 34 participants in each group.The study will be a double-blind randomized control trial. Patients will be recruited based on surgery type (hysteroscopy) and consented using a written consent by the research coordinator with sufficient time to ensure patient comprehension and allow for any questions. The consent process will happen in the pre-operative appointment. Participants will then be randomized to either the standard of care of 80mmHg or the experimental pressure of 60 mmHg for uterine filling pressure via an automated randomization program. The physician performing the surgery and the patient will not know what group they are assigned to. The procedure involved in the study will be hysteroscopy. Hysteroscopy is a procedure that is used to diagnose and sometimes treat intrauterine pathologies. In order to visualize the uterus, pressurized saline is used to distend the uterus.

In this study, the specific hysteroscopic procedure will involve the removal of uterine fibroids with a MyoSure Hysteroscopic Morcellator device. These tissue samples will be collected and sent to Pathology to be weighed. During the surgery, the surgeon will be able to request an adjustment pressure if visualization is not adequate. Physicians will start with a pressure of 80mmHg. Once physician is ready to introduce the myosure hysteroscopy device, the pressure level will then be randomized. During the procedure, monitoring will be done by anesthesia through the use of pulse oximetry and measurement of vitals during the Monitored Anesthesia Care. There is also real-time monitoring of hysteroscopic fluid deficit via the fluid management system that is attached to the hysteroscopic pump. Fluid deficit can also be confirmed by the nurse who manually counts the amount of fluid used during theprocedure. Per policy, once a 2500mL deficit is reached, the procedure is terminated. After the surgery, the surgeon will fill out a questionnaire that measures the outcomes of surgeon satisfaction and visualization during the procedure. The other end points of procedure time, specimen weight, volume of normal saline used, any changes in pressure needed during the surgery, and whether the patient required Lasix post-operatively will also be collected at this time.

ELIGIBILITY:
Inclusion Criteria:

* Patients electing for operative or diagnostic hysteroscopy procedures for management of polyps and fibroids
* Age equal to or greater than 18
* Ability to understand and willingness to sign consent form. We will include non-English speaking patients in this study

Exclusion Criteria:

* Patients electing for operative and diagnostic hysteroscopy procedures with polyps and fibroids
* Patients under the age of 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Physician Survey to assess visualization | Through study completion, an average of 1 year
  Determining whether lowering pressure on hysteroscopic morcellator during hysteroscopy, using block randomization, affects visualization for surgeon using a post-op survey for surgeon to gauge outcomes.
Procedure Time | Through study completion, an average of 1 year
  Duration of surgery to assess if pressure changes affects length of surgery time.
Specimen Weight | Through study completion, an average of 1 year
  Specimen will be sent to pathology to note weight in grams.
Amount of Fluid | Through study completion, an average of 1 year
  Volume of normal saline used during procedure.
Lasix administered post-operatively | Through study completion, an average of 1 year
  Noting yes or no if Lasix was administered post-operatively.
Change in pressure was needed | Through study completion, an average of 1 year
  Noting if pressure needed changing by surgeon during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Magdy P Milad, MD, MM, Principal Investigator — Northwestern University
Locations (1):
- Center for Comprehensive Gynecology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will only involve consent forms, which will be stored in a locked cabinet in the research coordinators office along with the updated protocol and other study materials. The survey for the surgeon performing the procedure will be stored in the same place and used for data analysis.

DOCUMENTS (2):
  • Study Protocol (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04550429/Prot_000.pdf
  • Informed Consent Form (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT04550429/ICF_001.pdf